CLINICAL TRIAL: NCT04018001
Title: Comparative Analysis of Adherence and Effectiveness Outcomes Between Rheumatoid Arthritis (RA) Patients Treated With Tofacitinib Modified Release (MR) Formulation 11mg Once Daily (QD) and Tofacitinib Immediate Release (IR) Formulation 5 mg Twice Daily (BID) Within a United States (US) Healthcare Claims Database
Brief Title: Comparative Analysis of Adherence and Effectiveness Outcomes Between Rheumatoid Arthritis (RA) Patients Treated With Tofacitinib Modified Release (MR)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921349
Record Dates: First submitted 2019-06-11; First posted 2019-07-12 (Actual); Results first posted 2020-04-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Truven Health MarketScan Research Database: individuals who are privately insured and with Medicare Supplemental insurance

SUMMARY:
The purpose of this study is to compare adherence, persistence, and effectiveness among patients initiating tofacitinib Modified Release (MR) with tofacitinib Immediate Release (IR).

ELIGIBILITY:
Inclusion Criteria:

* At least one claim for tofacitinib between 01 January 2014 and 31 January 2017 (the identification period).
* Presence of The International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9 CM) code for RA (in any position) during the one-year pre-index period or on the index date. ICD-9 = 714.0x-714.4x & 714.81 or ICD10 = M05.* & M06.0*-M06.3* or M06.8*-M06.9*.
* At least 18 years old as of the index date.

Exclusion Criteria:

* Patients with claims for other conditions for which biologics are used during the one-year pre-index period or on the index date: ankylosing spondylitis, Crohn's disease, psoriasis, psoriatic arthritis, or ulcerative colitis will be excluded from the study.
* Patients with evidence of the index medication during the one-year pre-index period will be removed from the analysis. Patients will be allowed to have been treated with other biologics approved for RA (Tumor-Necrosis Factor-alpha inhibitors (TNFi) [adalimumab (Humira), etanercept (Enbrel), certolizumab pegol (Cimzia), golimumab (Simponi), infliximab (Remicade)] and non-TNFi's with alternative mechanisms of action [abatacept (Orencia), and rituximab (Rituxan), anakinra (Kineret), tocilizumab (Actemra)]) during the one-year pre-index period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals initiating tofacitinib
Sampling Method: Non-Probability Sample
Enrollment: 1057 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cohen SB, Greenberg JD, Harnett J, Madsen A, Smith TW, Gruben D, Zhang R, Lukic T, Woolcott J, Dandreo KJ, Litman HJ, Blachley T, Lenihan A, Chen C, Rivas JL, Dougados M. Real-World Evidence to Contextualize Clinical Trial Results and Inform Regulatory Decisions: Tofacitinib Modified-Release Once-Daily vs Immediate-Release Twice-Daily for Rheumatoid Arthritis. Adv Ther. 2021 Jan;38(1):226-248. doi: 10.1007/s12325-020-01501-z. Epub 2020 Oct 9. PMID 33034006
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921349

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was a retrospective follow-up study of participants treated with index medication (tofacitinib) and enrolled in a health insurance plan for a minimum of 24 months.
Groups:
- Tofacitinib Modified Release (MR): Participants with Rheumatoid Arthritis (RA) who were treated with Tofacitinib 11 milligram (mg) MR tablet, orally, once daily, between 01 March 2016 and 31 October 2018 (identification period) and enrolled in a commercial or Medicare insurance plan for 1 year before the index date to at least 1 year after the index date, were included in this study. Index date was the date of first claim for 30-day supply of tofacitinib by participants to their insurance provider during identification period. Data collected retrospectively for participants included in this study.
- Tofacitinib Immediate Release (IR): Participants with RA who were treated with Tofacitinib 5 mg IR tablet orally, twice daily, between 01 March 2016 and 31 October 2018 and enrolled in a commercial or Medicare insurance plan for 1 year before the index date to at least 1 year after the index date, were included in this study. Index date was the date of first claim for 30-day supply of tofacitinib by participants to their insurance provider during identification period. Data collected retrospectively for participants included in this study.
Period: Overall Study
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Started | 678 | 379
Completed | 678 | 379
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR) | Total
Number analyzed (Participants) | 678 | 379 | 1057
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.35 (10.20) | 53.97 (10.91) | 54.22 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 556 | 311 | 867
  Male | 122 | 68 | 190
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Combination Therapy [Number; unit: participants] — Combination therapy was defined as first comedication with any Conventional synthetic disease-modifying antirheumatic drug (csDMARD).
  participants | 370 | 214 | 584
Use of non-steroidal antiinflammatory drug (NSAID)s Pre-Index [Number; unit: participants] — Participants who took NSAIDs before index date were reported.
  participants | 297 | 190 | 487
Number of Advanced Therapies At Index [Number; unit: advanced therapies] — Participants who took no advance therapy (0), 1 advance therapy (1) 2 advance therapies (2), and atleast 3 advance therapies (>=3) were reported.
  advanced therapies
    0 | 142 | 93 | 235
    1 | 240 | 128 | 368
    2 | 192 | 97 | 289
    >=3 | 104 | 61 | 165
Insurance type [Number; unit: participants]
  Commercial Claims and Encounters (CCAE) | 596 | 327 | 923
  Medicare (MDCR) | 82 | 52 | 134
Region [Number; unit: participants]
  North Central Region | 110 | 65 | 175
  Northeast Region | 125 | 74 | 199
  South Region | 371 | 191 | 562
  Unknown Region | 2 | 0 | 2
  West Region | 70 | 49 | 119
Year and month of the participant's index date [Number; unit: participants]
  2016-03 | 1 | 45 | 46
  2016-04 | 5 | 45 | 50
  2016-05 | 22 | 31 | 53
  2016-06 | 25 | 17 | 42
  2016-07 | 17 | 15 | 32
  2016-08 | 40 | 21 | 61
  2016-09 | 32 | 20 | 52
  2016-10 | 33 | 13 | 46
  2016-11 | 50 | 15 | 65
  2016-12 | 38 | 20 | 58
  2017-01 | 33 | 18 | 51
  2017-02 | 48 | 19 | 67
  2017-03 | 44 | 14 | 58
  2017-04 | 36 | 12 | 48
  2017-05 | 49 | 19 | 68
  2017-06 | 34 | 11 | 45
  2017-07 | 43 | 13 | 56
  2017-08 | 51 | 13 | 64
  2017-09 | 30 | 10 | 40
  2017-10 | 39 | 8 | 47
  2017-11 | 8 | 0 | 8
Index Medication [Number; unit: participants] — Participants who took index medication were reported.
  participants | 678 | 379 | 1057

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Met All Effectiveness Criteria up to 12 Months From the Index Date
Description: Effectiveness criteria: 1) High adherence with proportion of days covered greater than or equal to [>=] 0.8; 2) No increase in index medication dose; 3) No use of an advanced therapy other than index therapy 4) No addition/claims of conventional synthetic disease-modifying antirheumatic drug; 5) If no oral glucocorticoid prescriptions in the 6 months prior to index date, then no more than 30 total days supply of oral glucocorticoids between 3-12 months post index or if at least 1 claim for oral glucocorticoids during 6 months pre-index, then oral glucocorticoid not increased by >=20% between 6-12 months post-index compared to 6 months before index date (6) Participants have one or fewer glucocorticoid injections during 3-12 months after index date. Adherence was defined as percentage of time with medication on hand. Participants who met all 6 effectiveness criteria considered as treated effectively.
Time Frame: Up to 12 months from index date (Index date: date of first claim for tofacitinib by participants to insurance provider during identification period of 2.6 years)
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 33.33 | 25.86
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0115, Chi-squared
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0227, Regression, Logistic — To better assess true effect of treatment,analysis with participant's baseline characteristic was adjusted to remove influence on the outcome measure; Odds Ratio (OR) = 1.410198, 95% CI 2-sided [1.0492535 to 1.8953079]

2. Primary Outcome: Mean Treatment Persistence Duration for Tofacitinib up to 12 Months From Index Date
Description: Treatment persistence with tofacitinib was defined as participants who did not switch to another advanced therapy or discontinued tofacitinib. Discontinuation of tofacitinib was defined as at least 60 days gap between the run out of prior tofacitinib prescription and subsequent treatment. The run out date was the prescription fill date + day supply -1.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study. Here "Overall number of participants analyzed" signifies only those participants who had data available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 142 | 93
days | 243.4 (135.1) | 235.7 (129.6)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.3564, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.2629, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.9022, 95% CI 2-sided [0.7534 to 1.0803]

3. Primary Outcome: Mean Adherence to Tofacitinib by Medication Possession Ratio (MPR) up to 12 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with MPR >=0.8 were considered to show high adherence and participants with MPR less than (<) 0.8 were considered as low adherence. MPR was calculated as the total days supply of tofacitinib between the first and including the last tofacitinib prescription divided by the time between the first through and including last index therapy prescription days supply.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
ratio | 0.89 (0.15) | 0.86 (0.18)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0123, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0047, Generalized linear model — [p-value comment as in outcome 1, analysis 2]; Difference in Least Squares (LS) Means = 0.0300853, 95% CI 2-sided [0.0092322 to 0.0509385]

4. Primary Outcome: Percentage of Participants With Adherence to Tofacitinib as Assessed by Greater Than or Equal to (>=) 0.8 Medication Possession Ratio (MPR) up to 12 Months From the Index Date
Description: Adherence is defined as percentage of time with medication on hand. Participants with MPR >=0.8 were considered to show high adherence. MPR was calculated as the total days supply between the first and including the last tofacitinib prescription divided by the time between the first through and including last index therapy prescription days supply.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 80.09 | 69.92
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0002, Chi-squared
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.7910474, 95% CI 2-sided [1.3167136 to 2.4362554]

5. Primary Outcome: Mean Adherence to Tofacitinib by Proportion of Days Covered (PDC) up to 12 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with PDC >= 0.8 were considered to show high adherence and participants with PDC <0.8 were considered to show low adherence. PDC was defined as number of days covered by arrays for each fill or administration during the denominator periods of 360 days post-index.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
ratio | 0.63 (0.33) | 0.62 (0.30)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.4071, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.6143, Generalized linear model — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = 0.0104065, 95% CI 2-sided [-0.030062 to 0.0508746]

6. Primary Outcome: Primary: Percentage of Participants With Adherence to Tofacitinib as Assessed by Greater Than or Equal to (>=) 0.8 Proportion of Days Covered (PDC) up to 12 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with PDC >=0.8 were considered to show high adherence. PDC was defined as number of days covered by arrays for each fill or administration during the denominator periods of 360 days post-index.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 48.23 | 37.73
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0010, Chi-squared
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.5211586, 95% CI 2-sided [1.1594614 to 1.9956882]

7. Secondary Outcome: Mean Treatment Persistence Duration for Tofacitinib up to 6 Months From Index Date
Description: as for outcome 2
Time Frame: Up to 6 months from index date (Index date: date of first claim for tofacitinib made by participants to their insurance provider during identification period of 2.6 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
days | 143.7 (57.7576) | 146.3 (55.6362)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.4595, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.3354, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.1225, 95% CI 2-sided [0.8873 to 1.4201]

8. Secondary Outcome: Mean Adherence to Tofacitinib by Medication Possession Ratio (MPR) up to 6 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with MPR >=0.8 were considered to show high adherence and participants with MPR <0.8 were considered to show low adherence. MPR was calculated as the total days supply of tofacitinib between the first and including the last tofacitinib prescription divided by the time between the first through and including last index therapy prescription days supply.
Time Frame: as for outcome 7
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
ratio | 0.90 (0.14) | 0.88 (0.16)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.1130, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.1194, Generalized linear model — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = 0.0151242, 95% CI 2-sided [-0.003908 to 0.0341568]

9. Secondary Outcome: Percentage of Participants With Adherence to Tofacitinib as Assessed by Greater Than or Equal to (>=) 0.8 Medication Possession Ratio (MPR) up to 6 Months From the Index Date
Description: as for outcome 4
Time Frame: as for outcome 7
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 82.45 | 76.52
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0200, Chi-squared
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0364, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.4143816, 95% CI 2-sided [1.0221455 to 1.9571335]

10. Secondary Outcome: Mean Adherence to Tofacitinib by Proportion of Days Covered (PDC) up to 6 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with PDC >= 0.8 were considered to show high adherence and participants with PDC <0.8 were considered to show low adherence. PDC was defined as number of days covered by arrays for each fill or administration during the denominator periods of 180 days post-index.
Time Frame: as for outcome 7
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
ratio | 0.71 (0.28) | 0.71 (0.27)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.9031, t-test, 2 sided
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.6376, Generalized linear model — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -0.008587, 95% CI 2-sided [-0.044317 to 0.0271416]

11. Secondary Outcome: Percentage of Participants With Adherence to Tofacitinib as Assessed by Greater Than or Equal to (>=) 0.8 Proportion of Days Covered (PDC) up to 12 Months From the Index Date
Description: Adherence was defined as percentage of time with medication on hand. Participants with PDC >=0.8 were considered to show high adherence. PDC was defined as number of days covered by arrays for each fill or administration during the denominator periods of 180 days post-index.
Time Frame: as for outcome 7
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 56.49 | 53.56
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.3584, Chi-squared
Statistical Analysis 2: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.4510, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.1077385, 95% CI 2-sided [0.8489444 to 1.4454238]

12. Other Pre Specified Outcome: Percentage of Participants Who Showed Persistence for Tofacitinib up to 12 Months From the Index Date
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 51.62 | 45.65
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.0624, Chi-squared

13. Other Pre Specified Outcome: Percentage of Participants Who Showed Persistence for Tofacitinib up to 6 Months From the Index Date
Description: as for outcome 2
Time Frame: as for outcome 7
Population: Analysis was performed on all participants included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 678 | 379
percentage of participants | 68.14 | 70.18
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Test type: Superiority; p = 0.4914, Chi-squared

ADVERSE EVENTS:
Description: Due to the nature of claims data base from which these data where queried, no adverse events were collected in this study.
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT04018001/Prot_SAP_000.pdf